CLINICAL TRIAL: NCT02338895
Title: An Ultrasound- Guided Algorithm for the Management of Oliguria in Septic Shock
Brief Title: Algorithm for Oliguria in Septic Shock
Acronym: AMOSS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Principal Investigator, Nawal Salahuddin, Consultant Physician, King Faisal Specialist Hospital & Research Center
Other Study IDs: RAC # 2141039
Record Dates: First submitted 2015-01-11; First posted 2015-01-14 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Acute Kidney Injury
Keywords: acute kidney injury, oliguria,renal ultrasound
MeSH Terms: conditions — Acute Kidney Injury; Oliguria | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- acutly oliguric patients with ultrasound: Patients with septic shock and acute oliguria that will undergo bedside ultrasonographic assessment of inferior vena caval diameter, respiratory variation and renal perfusion.
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Ultrasound of inferior vena cava and kidneys

SUMMARY:
Acute Kidney Injury (AKI) develops in 88% to 30% of critically ill patients admitted to an intensive care unit and is a strong predictor of mortality.Therefore any management strategy that prevents progression of renal risk to injury or failure has the potential to improve outcomes in these patients.Conventional management of acute oliguria in shock has been to blindly 'push' fluids to improve renal perfusion or to give loop diuretics once fluid loading has been considered as accomplished. However both volume overload and 'blind' attempts at fluid removal can worsen renal injury and have been associated with higher mortality by venous overcongestion and inappropriate hypovolemia. It seems reasonable to assume that a bedside test to visualize volume status and renal perfusion may assist in improving outcomes in this cohort.The investigators developed a goal-directed ultrasonographic protocol to provide immediate hemodynamic information in acutely oliguric patients with shock as well as a management algorithm for guiding therapy. The investigators incorporated IVC diameter measurement, respiratory variation and response to a passive leg raise to assess whether further fluid boluses were required and a measurement of renal perfusion to determine whether diuretics or renal replacement therapy were indicated. The investigators aim to measure the effects of this management protocol on the rates of AKI in the study participants as compared to prior to the implementation of the protocol.The study design is a prospective, observational. Since this is a proof of concept study, the projected sample size is 40 patients. An interim analysis will be carried out after 20 patients are enrolled and a further 20 will be enrolled as necessary

DETAILED DESCRIPTION:
BACKGROUND & INTRODUCTION:

Acute Kidney Injury (AKI) develops in 88% to 30% of critically ill patients admitted to an intensive care unit. While AKI of any severity is a strong predictor of mortality (1-4), both morbidity and mortality increase with increasing severity of renal injury(2). Therefore any management strategy that prevents progression of renal risk to injury or failure has the potential to improve outcomes in these patients.

Conventional management of acute oliguria in shock has been to blindly 'push' fluids to improve renal perfusion or to give loop diuretics once fluid loading has been considered as accomplished. However both volume overload and 'blind' attempts at fluid removal can worsen renal injury and have been associated with higher mortality by venous overcongestion (5) and inappropriate hypovolemia (6-8). It seems reasonable to assume that a bedside test to visualize volume status and renal perfusion may assist in improving outcomes in this cohort. Intensive care unit (ICU) bedside ultrasound has become the standard of care for critically ill patients(9-18). In patients with shock, inferior vena cava ultrasonographic evaluation for 'fluid responsiveness' is routinely used to direct resuscitation (19-21) by direct measurement of IVC diameter and respiratory variation or by the response to a noninvasive fluid bolus from a passive leg raise (22). Doppler ultrasound of intrarenal vessels has also been described as a tool to assess renal perfusion (23-27).

The investigators developed a goal-directed ultrasonographic protocol to provide immediate hemodynamic information in acutely oliguric patients with shock as well as a management algorithm for guiding therapy. The investigators incorporated IVC diameter measurement, respiratory variation and response to a passive leg raise to assess whether further fluid boluses were required and a measurement of renal perfusion to determine whether diuretics or renal replacement therapy were indicated.

The objectives are to measure the effects of this management protocol on the rates of AKI in the study participants as compared to prior to the implementation of the protocol.

METHODS:

1. Study Design: Prospective, Observational 2. Study Patients:

* Inclusion criteria: Critically ill, adult patients AND with acute oliguric renal failure AND within 6 hours of presentation
* Exclusion criteria:

  i. Patients with pre-existing chronic renal failure ii. Patients on renal replacement therapy/ Dialysis iii. Patients with poor sonographic windows

  3. Variables to be measured:
* Dependent variables:

  a. Demographic identifiers; age, gender, comorbidity, admitting diagnosis, APACHE II scores, b. Renal perfusion as measured by color Doppler c. Daily fluid balance, d. Mean hourly urine output, e. Vasopressor use, f. Daily serum Creatinine g. Response to diuretics h. Dose of diuretic that resulted in urine output
* Outcome variables:

  1. Incidence of renal failure (classified into RIFLE categories; Risk, Injury, Failure, Loss of Function, End-Stage: see Appendix 1),
  2. ICU length of Stay,
  3. ICU mortality

Materials & Methodologies:

1. Screening & Enrollment of patients:

   1. All ICU patients admitted to the ICU will be screened for enrollment.
   2. Those meeting inclusion criteria will have their Demographic information entered in Case Record Forms (Appendix 2: Sample CRF)
   3. Ultrasound examinations will be carried out and results entered into the CRF.

      o For patients found to be intravascularly dehydrated (those with > 2 cm IVC diameter (IVCd) or >15% variation in IVCd or an increase of > 15% in IVCd with a passive leg raise maneuver), the results will be communicated to the managing ICU team for fluid resuscitation
      * For patients found to be adequately hydrated, renal perfusion will be assessed by observing flow in the interlobar and arcuate vessels by colour Doppler and the renal resistive index will be measured.
      * The results of no perfusion or perfusion present will be communicated to the managing ICU team for recommendation of high dose diuresis
2. Ultrasonographic assessment of Inferior Vena Cava Measurement of the inferior vena cava diameter, and respiratory variation by ultrasound (http://www.criticalecho.com/content/tutorial-4-volume-status-and-preload-responsiveness-assessment) Ultrasonographic assessment of the IVC will be done using a transthoracic, subcostal approach. The transducer will be positioned just below the xiphisternum 1-2cms to the right of the midline, with the marker dot pointing towards the sternal notch. After obtaining a 2-D image of the IVC entering the right atrium and verifying that the IVC visualization is not lost during movements of respiration, an M-mode line will be placed through the IVC 1 cm caudal from its junction with the hepatic vein, and an M-mode tracing obtained. This placement ensures that the intrathoracic IVC is not measured during any part of the respiratory cycle. The M-mode tracing will be recorded through 3- 4 respiratory cycles, the image frozen and using calipers, the maximum and minimum diameters of the IVC tracing measured. IVC variation will be quantified by measuring the difference between the maximum and minimum diameters on the M-mode tracing.

   Ultrasonographic assessment of Renal Perfusion by color Doppler

   Vessel localization and a semi-quantitative evaluation of renal perfusion will be carried out using the following staging method. (http://link.springer.com/chapter/10.1007%2F978-3-642-10286-8_31 - page-1)

   Stage Quality of Renal Perfusion by color Doppler 0 Unidentifiable vessels 1 Few vessels in vicinity of hilum 2 Hilar and intralobar vessels in most of renal parenchyma 3 Renal vessels identifiable until the arcuate arteries in the entire field of view
3. Statistical Methods:

   1. Sample size & Sampling: Consecutive admissions to the ICU will be enrolled. Since this is a proof of concept study, the projected sample size is 40 patients. An interim analysis will be carried out after 20 patients are enrolled and a further 20 will be enrolled as necessary
   2. Analysis: Categorical variables will be reported as proportions or percentages, continuous variables as means or medians. Differences between groups will be estimated using CHI2, student t test or Mann-Whitney U test, as appropriate. Rates of renal injury from historical controls will be compared to rates measured using t test for paired samples. A p value =0.05 will be considered significant. SPSS version 22.0 will be used for all analysis.

ETHICAL CONSIDERATIONS:

1. Informed Consent for ultrasonographic examination. The use of use of ultrasound for the assessment and management of critically ill patients in the ICU and emergency room is considered as standard of care and is routinely practiced in ICUs around the world. Since ultrasound evaluation has become incorporated into usual ICU practice, written consent is not required in its routine use. We therefore ask for a waiver of informed consent since we will not be performing any deviation from usual ICU care and our study is simply a collection of practice into a protocolized form.

   (Please see References 9-27)
2. Research Advisory Committee (RAC) Review This protocol will be reviewed and approved by the hospital Research Advisory committee responsible for oversight of the study.

2. Subject Confidentiality & Protection of Rights of Control Subjects All case record forms, reports and other records will be identified only by the Study Identification Number (SID) to maintain subject confidentiality. All records will be kept in a password-protected file. All computer entry and networking programs will be done using SIDs only.

3. Study Modification/Discontinuation The study may be modified or discontinued at any time by the primary investigators and or Research Advisory Committee as part of their duties to ensure that research subjects are protected.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill, adult patients AND with acute oliguric renal failure AND within 6 hours of presentation

Exclusion Criteria:

* i. Patients with pre-existing chronic renal failure ii. Patients on renal replacement therapy/ Dialysis iii. Patients with poor sonographic windows

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Critically ill patients with septic shock presenting with acute oliguria
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
acute Kidney Injury | 28 days

SECONDARY OUTCOMES:
mortality | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Iqbal Hussain, MD, Principal Investigator — King Faisal Specialist Hospital & Research Center; Ashraf Nadeem, MD, Principal Investigator — King Faisal Specialist Hospital & Research Center
Locations (1):
- King Faisal specialist Hospital & Research Center, Riyadh, Ar Riyadh, Saudi Arabia